CLINICAL TRIAL: NCT05448989
Title: Efficacy and Safety of 1% Atropine "5+3" Regimen in Children and Adolescents Controlling Myopia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021SQ001
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% atropine 5+3 (Experimental): Put the 1% atropine eye drops into the conjunctival sac, then close the eyes and press the nasolacrimal duct used for 5 consecutive nights in the first week of each month, one night per week in the 2nd, 3rd, and 4th weeks; after 3 months of monocular application, change to the contralateral eye Total treatment time 1 year
  Interventions: Drug: 1% atropine 5+3
- 1% atropine weekly (Placebo Comparator): Put the 1% atropine eye drops into the conjunctival sac, then close the eyes and press the nasolacrimal duct once a week in both eyes Total treatment time 1 year
  Interventions: Drug: 1% atropine 5+3

INTERVENTIONS:
Drug: 1% atropine 5+3 — A method for myopia control using high-concentration atropine

SUMMARY:
Studies have shown that atropine eye drops are effective in controlling myopia in children and adolescents. 1% atropine ophthalmic drug has obvious curative effect for controlling myopia, but its side effects such as photophobia and blurred vision limit its popularization and use. In the early stage, our research group used 1% atropine "5+3" myopia control program and 1% atropine alternate eye myopia control program. Retrospective clinical research data showed that it could significantly reduce side effects and improve use compliance, but there is currently no evidence from prospective clinical studies.

DETAILED DESCRIPTION:
Studies have shown that atropine eye drops are effective in controlling myopia in children and adolescents. Among them, low-concentration atropine has few side effects and is the primary recommendation, but many clinical practices and studies suggest that its effect in controlling myopia is limited. 1% atropine ophthalmic drug has obvious curative effect advantages in controlling myopia, but its side effects such as photophobia and blurred vision limit its popularization and use. In the early stage, our research group used 1% atropine "5+3" myopia control (eye instillation for 5 consecutive nights in the first week of each month, one night per week in the 2nd, 3rd, and 4th weeks; after 3 months of monocular application, change to the contralateral eye), data from retrospective clinical studies have shown that it can significantly reduce side effects and improve compliance, but there is currently a lack of evidence from prospective clinical studies. Therefore, this study intends to use a randomized controlled trial, with 1% atropine used in both eyes once a week as the control group, to evaluate the effect of the "5+3" regimen in controlling myopia (spherical equivalent and axial length), safety (accommodation amplitude, amount of phoria, binocular vision function, etc.), and the compliance and side effects (photophobia, blurred vision, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years old;
* Both eyes are in line with the diagnosis of myopic refractive error and 0.25D < myopia spherical lens <4.00D after mydriasis, astigmatism <2.00D, binocular anisometropia <3.00D, and the best corrected distance vision is at least 0.8, myopia The force is at least 0.8;
* Visual function: Timus≤100 seconds, exophoria <5△, accommodation amplitude (AMP) ≥ age-related minimum accommodation amplitude value (minimum accommodation amplitude=15-0.25×age);
* No contraindications for atropine treatment such as acute eye inflammation, dry eye, keratoconus, diabetes, etc.;
* The written informed consent of the guardian and the child himself.

Exclusion Criteria:

* History of photosensitivity, glaucoma, blue eye syndrome, ocular hypertension, fundus macular lesions or damage;
* Corneal curvature examination, the average K value of the anterior surface of the cornea is ≥45;
* Patients with ocular trauma, oblique or surgical eyes, atopic keratoconjunctivitis and other chronic eye diseases;
* Those with previous ophthalmia, severe angular, conjunctival infection and other eye diseases;
* Patients with neurological diseases and allergic or contraindications to atropine or other therapeutic drugs;
* Received other treatments to control the development of myopia in the past, such as the use of anticholinergic drugs such as atropine within 3 months, or participated in other relevant researchers such as functional frame mirrors and multifocal flexible mirrors;
* Other circumstances judged by the investigator to be unsuitable to participate in the research.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent | Before atropine treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | 1months after treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | 3months after treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | 6months after treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | 9months after treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | 12months after treatment
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
axial length | Before atropine treatment
  axial length(AL), millimeter(mm), measured by IOL master
axial length | 1months after treatment
  axial length(AL), millimeter(mm), measured by IOL master
axial length | 3months after treatment
  axial length(AL), millimeter(mm), measured by IOL master
axial length | 6months after treatment
  axial length(AL), millimeter(mm), measured by IOL master
axial length | 9months after treatment
  axial length(AL), millimeter(mm), measured by IOL master
axial length | 12months after treatment
  axial length(AL), millimeter(mm), measured by IOL master

SECONDARY OUTCOMES:
accommodation amplitude | Before atropine treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
accommodation amplitude | 1months after treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
accommodation amplitude | 3months after treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
accommodation amplitude | 6months after treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
accommodation amplitude | 9months after treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
accommodation amplitude | 12months after treatment
  Accommodation amplitude is measured by the amount of diopter change as the target is moved closer, diopter(D)
amount of phoria | Before atropine treatment
  measured by Von-Graefe method, degree(°)
amount of phoria | 1months after treatment
  measured by Von-Graefe method, degree(°)
amount of phoria | 3months after treatment
  measured by Von-Graefe method, degree(°)
amount of phoria | 6months after treatment
  measured by Von-Graefe method, degree(°)
amount of phoria | 9months after treatment
  measured by Von-Graefe method, degree(°)
amount of phoria | 12months after treatment
  measured by Von-Graefe method, degree(°)
binocular vision function | Before atropine treatment
  measured by Titmus method, second
binocular vision function | 1months after treatment
  measured by Titmus method, second
binocular vision function | 3months after treatment
  measured by Titmus method, second
binocular vision function | 6months after treatment
  measured by Titmus method, second
binocular vision function | 9months after treatment
  measured by Titmus method, second
binocular vision function | 12months after treatment
  measured by Titmus method, second
photophobia | 1months after treatment
  the prevalence of photophobia known from Atropine Use and Adverse Reactions Questionnaire
photophobia | 3months after treatment
  the prevalence of photophobia known from Atropine Use and Adverse Reactions Questionnaire
photophobia | 6months after treatment
  the prevalence of photophobia known from Atropine Use and Adverse Reactions Questionnaire
photophobia | 9months after treatment
  the prevalence of photophobia known from Atropine Use and Adverse Reactions Questionnaire
photophobia | 12months after treatment
  the prevalence of photophobia known from Atropine Use and Adverse Reactions Questionnaire
blurred vision | 1months after treatment
  the prevalence of blurred vision known from Atropine Use and Adverse Reactions Questionnaire
blurred vision | 3months after treatment
  the prevalence of blurred vision known from Atropine Use and Adverse Reactions Questionnaire
blurred vision | 6months after treatment
  the prevalence of blurred vision known from Atropine Use and Adverse Reactions Questionnaire
blurred vision | 9months after treatment
  the prevalence of blurred vision known from Atropine Use and Adverse Reactions Questionnaire
blurred vision | 12months after treatment
  the prevalence of blurred vision known from Atropine Use and Adverse Reactions Questionnaire
Other discomfort | 1months after treatment
  Other discomfort reported by the patient but not included in the Atropine Use and Adverse Reactions Questionnaire
Other discomfort | 3months after treatment
  Other discomfort reported by the patient but not included in the Atropine Use and Adverse Reactions Questionnaire
Other discomfort | 6months after treatment
  Other discomfort reported by the patient but not included in the Atropine Use and Adverse Reactions Questionnaire
Other discomfort | 9months after treatment
  Other discomfort reported by the patient but not included in the Atropine Use and Adverse Reactions Questionnaire
Other discomfort | 12months after treatment
  Other discomfort reported by the patient but not included in the Atropine Use and Adverse Reactions Questionnaire

OTHER OUTCOMES:
lens thickness | Before atropine treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | 1months after treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | 3months after treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | 6months after treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | 9months after treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | 12months after treatment
  lens thickness(LT), millimeter(mm), measured by IOL master
lens power | Before atropine treatment
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | 1months after treatment
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | 3months after treatment
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | 6months after treatment
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | 9months after treatment
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | 12months after treatment
  lens power(LP), diopter(D), calculated by Bennett formula
anterior chamber depth | Before atropine treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
anterior chamber depth | 1months after treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
anterior chamber depth | 3months after treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
anterior chamber depth | 6months after treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
anterior chamber depth | 9months after treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
anterior chamber depth | 12months after treatment
  anterior chamber depth(ACD), millimeter(mm), measured by IOL master
corneal power | Before atropine treatment
  corneal power, diopter(D), measured by IOL master
corneal power | 1months after treatment
  corneal power, diopter(D), measured by IOL master
corneal power | 3months after treatment
  corneal power, diopter(D), measured by IOL master
corneal power | 6months after treatment
  corneal power, diopter(D), measured by IOL master
corneal power | 9months after treatment
  corneal power, diopter(D), measured by IOL master
corneal power | 12months after treatment
  corneal power, diopter(D), measured by IOL master
central corneal thickness | Before atropine treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
central corneal thickness | 1months after treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
central corneal thickness | 3months after treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
central corneal thickness | 6months after treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
central corneal thickness | 9months after treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
central corneal thickness | 12months after treatment
  central corneal thickness(CTC), micron(um), measured by IOL master
retinal thickness | Before atropine treatment
  retina thickness, microns(um), measured by SSOCT
retinal thickness | 1months after treatment
  retina thickness, microns(um), measured by SSOCT
retinal thickness | 3months after treatment
  retina thickness, microns(um), measured by SSOCT
retinal thickness | 6months after treatment
  retina thickness, microns(um), measured by SSOCT
retinal thickness | 9months after treatment
  retina thickness, microns(um), measured by SSOCT
retinal thickness | 12months after treatment
  retina thickness, microns(um), measured by SSOCT
choroidal thickness | Before atropine treatment
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | 1months after treatment
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | 3months after treatment
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | 6months after treatment
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | 9months after treatment
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | 12months after treatment
  choroidal thickness, microns(um), measured by SSOCT
ciliary muscle thickness | Before atropine treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary muscle thickness | 1months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary muscle thickness | 3months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary muscle thickness | 6months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary muscle thickness | 9months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary muscle thickness | 12months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | Before atropine treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | 1months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | 3months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | 6months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | 9months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | 12months after treatment
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xu, M.D., Study Director — Shanghai Eye Diseases Prevention Treatment Center
Locations (1):
- Shanghai Eye Diseases Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT05448989/Prot_000.pdf